CLINICAL TRIAL: NCT00001135
Title: A Phase III Randomized, Double-Blinded Study of Nevirapine for the Prevention of Maternal-Fetal Transmission in Pregnant HIV-Infected Women
Brief Title: A Study of Nevirapine to Prevent HIV Transmission From Mothers to Their Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: ACTG 316B; 11292 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2000-01-23; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Placebos; Pregnancy; Pregnancy Complications, Infectious; Nevirapine; Disease Transmission, Vertical; Labor; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
The purpose of this study is to see if giving the anti-HIV drug nevirapine (NVP) to HIV-positive pregnant women and their infants can help reduce the chance that a mother will give HIV to her baby during delivery.

NVP is a promising medication for blocking HIV transmission from HIV-positive mothers to their infants. NVP is inexpensive and is easily absorbed by the mother and transferred to the infant. It is thought that even a single dose to the mother and infant may provide enough protection to the baby during the time of exposure to HIV at birth.

DETAILED DESCRIPTION:
NVP has several properties that make it an attractive candidate for antiretroviral therapy to interrupt HIV-1 transmission in the intrapartum and early postpartum period. The pharmacokinetic profile suggests that NVP would be rapidly absorbed by the mother and transferred to the infant in utero when given during labor and delivery. The HIV-1 antiviral activity is rapid with significant reduction in plasma virus occurring within a few days of drug administration. In addition, NVP has been shown to penetrate cell-free virions and inactivate virion-associated reverse transcriptase (RT) in situ. This property would be potentially useful in inactivating cell-free virions in the genital tract as well as in breast milk. These characteristics of NVP suggest that treatment of an HIV-infected pregnant woman in labor with an oral dose of NVP may provide a prophylactic level of NVP in the infant during the time of exposure to virus in the birth canal and/or in the maternal blood. In addition, NVP may inactivate the virion-associated RT present in cell-free virions in the genital tract or breast milk.

Mothers are randomized to receive either a single oral dose of NVP during labor or the corresponding NVP placebo. Randomization occurs at any time after the 28th week of gestation. To assure balance between the treatment groups, the randomization is stratified using 2 factors: (1) antiretroviral therapy during the current pregnancy (no antiretroviral therapy at all, monotherapy [with no multi-agent therapy] for any duration, or multi-agent therapy for any duration), and (2) CD4 cell count at the time of randomization (less than 200 cells, 200 to 399 cells, or 400 cells or greater). Mothers are followed on-study for 4 to 6 weeks postpartum. All mothers are required to incorporate zidovudine (ZDV) into their current treatment regimen and should continue ZDV during delivery and give ZDV to their infants as recommended. ZDV will not be provided as part of the study.

Infants receive a single oral dose of NVP (or the corresponding placebo) administered between 48 and 72 hours of life. The infant's study drug is the same as the mother's randomized treatment assignment. Infants are dosed with study drug according to their randomization group regardless of whether the mother received study drug or not. Infants are followed for 6 months of life and are tested for HIV at birth, 4 to 6 weeks of life, 3 months of life, and 6 months of life.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are an HIV-positive pregnant woman.
* Have been pregnant for at least 28 weeks.
* Are at least 13 years of age (consent of parent or guardian is required if under 18).

Exclusion Criteria

You will not be eligible for this study if:

* You intend to breast-feed.
* You are allergic to benzodiazepines (a type of tranquilizer).
* You have a liver disorder.
* You have received nonnucleoside reverse transcriptase inhibitors (NNRTIs), a class of anti-HIV drugs.
* You refuse to take ZDV.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2009
Dates: Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorenbaum A, Study Chair; Sullivan JL, Study Chair
Locations (20):
- United States (19):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Univ of Miami (Pediatric), Miami, Florida
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan, Puerto Rico

REFERENCES:
- [Background] Cunningham CK, Balasubramanian R, Delke I, Maupin R, Mofenson L, Dorenbaum A, Sullivan JL, Gonzalez-Garcia A, Thorpe E, Rathore M, Gelber RD. The impact of race/ethnicity on mother-to-child HIV transmission in the United States in Pediatric AIDS Clinical Trials Group Protocol 316. J Acquir Immune Defic Syndr. 2004 Jul 1;36(3):800-7. doi: 10.1097/00126334-200407010-00006. PMID 15213563
- [Background] Watts DH, Balasubramanian R, Maupin RT Jr, Delke I, Dorenbaum A, Fiore S, Newell ML, Delfraissy JF, Gelber RD, Mofenson LM, Culnane M, Cunningham CK; PACTG 316 Study Team. Maternal toxicity and pregnancy complications in human immunodeficiency virus-infected women receiving antiretroviral therapy: PACTG 316. Am J Obstet Gynecol. 2004 Feb;190(2):506-16. doi: 10.1016/j.ajog.2003.07.018. PMID 14981398